CLINICAL TRIAL: NCT04501627
Title: A Multi-center, Single-arm, Prospective, Non-interventional Study on Vonoprazan in the Real-world Clinical Practice in China
Brief Title: A Study on Vonoprazan in the Real-world Clinical Practice in China
Acronym: VIEW
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vonoprazan-4007
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Esophagitis Peptic
Keywords: Drug Therapy
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with RE: Participants diagnosed with RE who have received 20 milligram (mg) of vonoprazan in routine clinical practice, will be observed prospectively. Data will be collected from participants' medical records, self-reported questionnaires and recorded information on symptom via diaries.

SUMMARY:
The purpose of this study is to evaluate the safety of Vonoprazan by assessing all adverse events (AEs), serious adverse events (SAEs), and adverse drug reactions (ADRs) in routine clinical settings in China.

DETAILED DESCRIPTION:
This is a prospective, non-interventional study in Chinese participants with RE who are receiving or will receive the standard treatment of vonoprazan. This study will assess the safety and effectiveness of vonoprazan in the real-world clinical practice.

The study will enroll approximately 3000 participants. The data will be collected through participants' medical records, self-reported questionnaires, and recorded information on symptom via diaries. All the participants will be assigned to a single observational cohort:

• Participants with RE

The multi-center trial will be conducted in China. The standard treatment will be of 4 weeks or it may reach up to 8 weeks if the dosing proves insufficient. All participants will be followed up for additional 2 weeks after the standard treatment. The overall duration of the study will be approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Must be undergoing treatment with Vonoprazan.
2. Must be at least 18 years old.
3. Provide signed informed consent indicating that they (or a legally acceptable representative) have been informed of all pertinent aspects of the study and are willing to participate.

Exclusion Criteria:

1. Are currently enrolled in or plan to participate in any other clinical trials (that is interventional study).
2. Are contraindicated for Vonoprazan according to Product Package Insert.
3. With a known hepatic function impairment, including jaundice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese participants who are prescribed with vonoprazan treatment in real-world clinical practice will be observed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Reporting one or More AEs | Up to Week 10
Percentage of Participants Reporting one or More SAEs | Up to Week 10
Percentage of Participants Reporting one or More ADRs | Up to Week 10
  ADRs refers to AE related to administered drug.

SECONDARY OUTCOMES:
Percentage of Participants with Endoscopic Healing of Reflux Esophagitis (RE) During 4-week Treatment | Baseline up to Week 4
  Endoscopic healing is defined as participants endoscopically diagnosed as Los Angeles classification Grade O during the treatment phase. The definitions of each grade are: Grade O (No mucosal break), Grade A (Mucosal break less than [<] 5 millimeter [mm]), Grade B (Mucosal break greater than or equal to [>=] 5 mm), Grade C (Mucosal break continuous between two or more folds and <75% of the esophageal circumference) and Grade D (Mucosal break >=75 percent [%] of the esophageal circumference).
Percentage of Participants with Endoscopic Healing of RE During 8-week Treatment | Baseline up to Week 8
  Endoscopic healing is defined as participants endoscopically diagnosed as Los Angeles classification Grade O during the treatment phase. The definitions of each grade are: Grade O (No mucosal break), Grade A (Mucosal break <5 mm), Grade B (Mucosal break >=5 mm), Grade C (Mucosal break continuous between two or more folds and <75% of the esophageal circumference) and Grade D (Mucosal break >=75% of the esophageal circumference).
Percentage of RE Participants Without Gastroesophageal Reflux Disease (GERD) Typical Symptoms | Baseline and Week 4
  The severity of participants' GERD symptoms based on the investigator's assessment among all participants will be evaluated at Baseline and Week 4. GERD symptoms will be assessed on a 5-point scale, wherein 1= no symptom, 2= mild, 3= moderate, 4= severe and 5= very severe. GERD symptoms include heartburn (HB), acid regurgitation (AR), dysphagia (dysp), belching (bch) and epigastric pain (EP). The participants without any GERD typical symptoms will be analyzed.
Percentage of Participants With Heartburn at Baseline Achieving Complete Heartburn Symptom Relief During the First Week of Treatment | Baseline up to Week 1
  The complete relief of heartburn symptom is defined as no such symptom occurred on 7 consecutive days. Percentage of participants with complete relief during Week 1 will be reported. Reported data will be the percentage of participants, calculated by the (number of participants with complete heartburn symptom relief) divided by (the total number of participants) *100%.
Percentage of Participants with Night Time Heartburn at Baseline Achieving Complete Night Time Heartburn Symptom Relief During the First Week of Treatment | Baseline up to Week 1
  The complete relief of night time heartburn symptoms is defined as no such symptom occurred on 7 consecutive nights. Percentage of participants with complete relief during Week 1 will be reported. Reported data will be the percentage of participants, calculated by the (number of participants with complete night time heartburn symptom relief) divided by (the total number of participants) *100%.
Percentage of Participants With Acid Regurgitation at Baseline Achieving Complete Acid Regurgitation Symptom Relief During the First Week of Treatment | Baseline up to Week 1
  The complete relief of acid regurgitation symptom is defined as no symptoms of acid regurgitation occurring on 7 consecutive days. Percentage of participants with complete relief during Week 1 will be reported. Reported data will be the percentage of participants, calculated by the (number of participants with complete acid regurgitation symptom relief) divided by (the total number of participants) *100%.
Percentage of Participants With Night Time Acid Regurgitation Symptom at Baseline Achieving Complete Night Time Acid Regurgitation Symptom Relief During the First Week of Treatment | Baseline up to Week 1
  The complete relief of acid regurgitation symptoms durng night time is defined as no symptoms of acid regurgitation occurring on 7 consecutive nights. Percentage of participants with complete relief during Week 1 will be reported. Reported data will be the percentage of participants, calculated by the (number of participants with complete night time acid regurgitation symptom relief) divided by (the total number of participants) *100%.
Change from Baseline in Gastroesophageal Reflux Disease Questionnaire (GerdQ) Score at Week 4 | Baseline up to Week 4
  GerdQ is a self-completed participant questionnaire that is used to assess whether the following symptoms of RE are improved under treatment: heartburn, regurgitation, stomach pain, nausea, sleep disturbance and use of additional medication due to heartburn/regurgitation. Symptom frequency will be assessed for the week passed using following answers: 0 days, 1 day, 2-3 days, and 4-7 days. Each answer will be assigned a score from 0 to 3 (heartburn, regurgitation, sleep disturbance and use of additional medication due to heartburn/regurgitation) or from 3 to 0 (stomach pain, nausea). Total score will be calculated as a sum of 6 individual scores. GerdQ score was calculated as sum of these scores, giving a total score ranging from 0 to 18. When GerdQ >=8, the participants could be symptom based diagnosed as GERD. Total score of 0 to 2 points= 0% likelihood of GERD; 3 to 7 points= 50% likelihood of GERD; 8 to 10 points= 79% likelihood of GERD; 11 to 18 points= 89% likelihood of GERD.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (40):
- China (40):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Yongchuan Hospital of Chongqing Medical University, Yongchuan, Chongqing Municipality
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - Heilongjiang Provincial Hospital (Nanshang), Harbin, Heilongjiang
  - Henan Provincial Peoples Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Changshu No.2 People's Hospital, Changshu, Jiangsu
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Yantai Affiliated Hospital of Binzhou Medical College, Yantai, Shandong
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - General Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Affiliated Hospital of Medical School of Ningbo University, Ningbo, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - The Fourth Affiliated Hospital Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f9293e2296beb001e63bf63?idFilter=%5B%22Vonoprazan-4007%22%5D